CLINICAL TRIAL: NCT02547727
Title: Humoral and Cell-mediated Immune Responses After a Four-site Intradermal Rabies Booster Vaccination in Previously Rabies Immunized HIV-infected Adults
Brief Title: Immune Responses After a Four-site Intradermal Rabies Booster Vaccination in HIV-infected Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Saovabha Memorial Institute (Other)
Collaborators: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Suda Sibunruang, Principal investigator, Queen Saovabha Memorial Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 495/2015
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Rabies
Keywords: rabies vaccination
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Four-site intradermal vaccination (Experimental): 0.1 ml of rabies vaccine is distributed to 4 sites over both arms and thigh intradermally on day 0. Blood would be drawn for rabies neutralizing antibody, OX-40 assay and cytokines assessment on day 0,7,14.
  Interventions: Biological: rabies vaccine
- Intramuscular vaccination (Active Comparator): 0.5 ml of rabies vaccine is injected to one arm on day 0 and 3.Blood would be drawn for rabies neutralizing antibody, OX-40 assay and cytokines assessment on day 0,7,14.
  Interventions: Biological: rabies vaccine

INTERVENTIONS:
Biological: rabies vaccine — Rabies vaccine is injected according to the protocol then blood would be drawn for rabies neutralizing antibody, OX-40 assay and cytokines assessment on day 0,7,14.

SUMMARY:
A four-site intradermal rabies booster vaccination in HIV - infected patients who have ever received primary rabies vaccination could improve their immune response to this kind of vaccine.

DETAILED DESCRIPTION:
A four-site intradermal rabies booster vaccination has shown higher immune response than conventional intramuscular rabies booster vaccination in healthy persons. So, the investigators hypothesized the same outcome in HIV - infected patients.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected patients
* Age 18 - 60 years
* Received primary rabies immunization

Exclusion Criteria:

* Have any active opportunistic infections
* Received blood or blood product within 3 months
* Allergy to vaccine or any vaccine components
* Received anti-malarial drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Rabies neutralizing antibody titers | Change from baseline of geometric mean titres of rabies neutralizing antibody titres at 2 weeks
  Rabies neutralizing antibody titers would be represented and compared by geometric mean titers (GMTs)

SECONDARY OUTCOMES:
Specific T cell response | Change from baseline of percentages of rabies-antigen specific CD4+ T cells at 2 weeks
  Specific T cell response is measured by OX-40 assay
Cytokines assessment | Change from baseline of cytokines levels at 1 week
  A few cytokines levels are measured by multiplex bead array assay

CONTACTS AND LOCATIONS:
Overall Officials: Suda Sibunruang, MD, Principal Investigator — Queen Saovabha Memorial Institute. Faculty of Medicine, Chulalongkorn university
Locations (1):
- Queen Saovabha Memorial Institute, Thai Red Cross Society, Bangkok, Thailand